CLINICAL TRIAL: NCT05776212
Title: Quantitative-imaging in Cardiac Transthyretin Amyloidosis
Acronym: I-CARE
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); Netherlands Heart Foundation (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Other Study IDs: 202000469; 2020-003350-72 (EudraCT Number)
Record Dates: First submitted 2023-01-26; First posted 2023-03-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: ATTR-CM
Keywords: Amyloidosis; Heart failure; 18F-fluoride positron emission tomography (PET); Cardiovascular magnetic resonance (CMR); Tafamidis
MeSH Terms: conditions — Amyloidosis; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Work package 1 - Optimisation of 18F-fluoride PET in ATTR-CM: Optimise 18F-fluoride PET imaging of ATTR-CM with increased myocardial tissue to background ratio (TBR) uptake values to provide a state-of-the-art imaging modality for use in the other work packages. (n=15, ATTR-CM subjects)
  Interventions: Radiation: 18F-fluoride PET
- Work package 2 - Differentiation ATTR-CM from phenocopies: Establish the optimised 18F-fluoride TBR threshold that best differentiates ATTR-CM (n=100) from phenocopies (subjects with light chain amyloidosis, n=20 and subjects with hypertrophic cardiomyopathy, n=20).
  Interventions: Radiation: 18F-fluoride PET
- Work package 3 - In vivo calibration of 18F-fluoride PET: In vivo calibration of 18F-fluoride PET as a marker of the myocardial ATTR burden, calibrating optimised TBR values against the current imaging standard cardiac magnetic resonance imaging extracellular volume. (Subjects with ATTR-CM, n=100)
  Interventions: Radiation: 18F-fluoride PET
- Work package 4 - Disease progression and treatment response: Establish ability of 18F-fluoride PET to track disease progression and treatment response in ATTR-CM at one year follow up. (Subjects with ATTR-CM, n=100)
  Interventions: Radiation: 18F-fluoride PET

INTERVENTIONS:
Radiation: 18F-fluoride PET — Positron emission tomography using 18F-fluoride as a tracer

SUMMARY:
Transthyretin amyloid cardiomyopathy (ATTR-CM), is a heart muscle disease that's stops the heart muscle working properly. With an ageing population, it is increasingly common but untreated, it has a poor prognosis. Several novel expensive treatments have become available, although we do not understand exactly how they work and why some patients respond, and others do not. The challenge is to develop better methods for monitoring the effects of these treatments, maximizing their benefits and cost-effectiveness. In I-CARE we aim to bring a new imaging technique, named 18F-fluoride PET, to the clinic and thereby improve the care of patients with ATTR-CM.

Hypotheses:

1. A delayed imaging protocol and state-of-the-art PET motion correction will optimise 18F-fluoride imaging in ATTR-CM and provide a clear threshold in myocardial TBR values for the diagnosis of ATTR-CM.
2. Optimised 18F-fluoride PET will provide a quantitative marker of the ATTR-CM burden that will allow disease progression and treatment response to be tracked.
3. Myocardial 18F-fluoride TBR values will reduce in patients responding to tafamidis treatment and increase in non-responders and patients not receiving therapy

DETAILED DESCRIPTION:
Studies have shown that there is calcium deposition in the heart muscle in ATTR-CM but exactly how this happens is not completely understood. Tafamidis, a new drug treatment, has shown improved outcomes for patients with ATTRCM by reducing hospitalisations and improving survival but the mechanism of action of Tafamidis is also not clearly understood yet. 18F-Fluoride PET/CT offers the opportunity to study this phenomenon of calcium deposition in ATTR-CM in more detail and study and track response to the new drug treatment. This will also provide an opportunity to investigate whether tafamidis therapy reduces calcium deposition in the heart muscle associated with ATTR-CM.

We have designed the study specifically to answer our research questions as best as possible, whilst keeping burdens to the patients at a minimum.

To the best of our knowledge this will be the first human study to utilise this imaging technique to assess and track response to the new drug treatment in ATTR-CM. We hope that it will provide major insights in to complex interactions at play, that could drive forward the development of novel therapeutic strategies for patients with ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

* Completion of informed consent
* Age > 40 years for patients with ATTR or AL cardiac amyloidosis and age >30 years for patients with HCM
* ATTR cardiac amyloid according to Expert Consensus Recommendations
* AL amyloidosis according to Expert Consensus Recommendations
* Hypertrophic cardiomyopathy according to European Society of Cardiology guidelines

Exclusion Criteria:

* Inability or unwilling to give informed consent
* Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial.
* Renal dysfunction (eGFR ≤30 mL/min/1.73m2)
* NYHA Class IV heart failure
* Patients with atrial fibrillation and poor rate control.
* Contraindications to MR
* Previous history of contrast allergy of adverse reactions (gadolinium)
* Contraindications to tafamidis therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with cardiac transthyretin amyloid
  * Patients with cardiac light chain amyloid
  * Patients with hypertrophic cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
TBR threshold | 1.5 years
  Tissue to background ratio with a good specificity and sensitivity to differentiatie subjects with ATTR-CM from subjects with phenocopies.

SECONDARY OUTCOMES:
Change in TBR | 2.5 years
  Change in TBR on 18F-fluoride PET/CT during one year of follow up.
Change in cardiac indices on CMR | 2.5 years
  Change in cardiac indices on magnetic resonance imaging, such as left ventricular ejection fraction
Change in cardiac biomarkers | 2.5 years
  Change in NT-ProBNP during one year of follow up.
Change in clinical measures | 2.5 years
  Change in clinical measures such as 6-minute walk test
TBR threshold | 6 months
  Specificity and sensitivity of TBR thresholds at different scanning times.
Change in Cardiac biomarkers | 2.5 years
  Change in cardiac high sensitivity troponin I during 1 year of follow up
Change in clinical measures | 2.5 years
  Change in KCCQ score during 1 year of follow up
Change in cardiac indices on CMR | 2.5 years
  change in left ventricular mass at 1 year follow up
Change in cardiac indices on CMR | 2.5 years
  change in extracellular volume at 1 year follow up
Change in cardiac indices on CMR | 2.5 years
  Change in left ventricular global longitudinal strain at 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dweck, MD PhD, Principal Investigator — Centre of Cardiovascular Science; Fabien Siepen, MD PhD, Principal Investigator — Heidelberg University
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication of the results in a peer-reviewed manuscript, the minimal data set underlying the findings will be made publicly available, either as part of the submission or through a stable, public repository such as EASY (DANS), DataverseNL or Zenodo. The "minimal data set" consists of the data set used to reach the conclusions drawn in the manuscript with related metadata and methods, and any additional data required to replicate the reported study findings in their entirety, including the values behind the means, standard deviations, and other measures reported, the values used to build graphs, and the points extracted from images for analysis. To obtain access to the full data set, a research proposal and analysis plan has to be submitted.

REFERENCES:
- [Derived] Tubben A, Prakken NHJ, Ivashchenko OV, Tingen HSA, Glaudemans AWJM, Noordzij W, Nienhuis HLA, van der Meer P, Slart RHJA. Feasibility of the absolute quantification and left ventricular segmentation of cardiac sympathetic innervation in wild-type transthyretin amyloidosis cardiomyopathy with [123I]-MIBG SPECT/CT: The I-NERVE study. J Nucl Cardiol. 2025 Mar;45:102146. doi: 10.1016/j.nuclcard.2025.102146. Epub 2025 Feb 3. PMID 39909199